CLINICAL TRIAL: NCT03133247
Title: A Phase 1, Open-Label, Multicenter, Non-Randomized, Dose Escalation Study to Evaluate the Safety and Tolerability of SHR-1316 in Subjects With Advanced Solid Tumors
Brief Title: A Trial to Evaluate Safety and Tolerability of SHR-1316 in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR1316-002
Record Dates: First submitted 2017-04-08; First posted 2017-04-28 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SHR-1316 dose-escalation (Experimental): SHR-1316 doses will be escalated sequentially in 5 cohorts.
  Interventions: Drug: SHR-1316

INTERVENTIONS:
Drug: SHR-1316 — PD-L1
  Other Names: HTI-1088

SUMMARY:
In many types of human tumors, PD-L1 is highly expressed. Such high expression has often been associated with poor prognosis in cancer patients. SHR-1316 is a humanized IgG4 monoclonal antibody that binds specifically to human PD-L1.

DETAILED DESCRIPTION:
This is a two-part, open-label, multicenter, non-randomized, dose escalation, Phase I study of repeated doses of SHR-1316 in subjects with advanced or metastatic solid tumors who have failed current standard anti-tumor therapies.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this study, each subject must meet all of the following criteria:

1. Male or female ≥18 years of age;
2. Diagnosed (histologically or cytologically) with solid tumors and documented as advanced or metastatic disease for which there is no known effective anti-tumor treatment (refractory to or relapsed from standard therapies). Subjects must have confirmation of this diagnosis through study-site analysis of fresh or archived tissue;
3. Failed no more than 1 prior PD-1/PD-L1 therapy and that more than 4 weeks has elapsed.
4. No prior cancer therapy within last 4 weeks;
5. ECOG Performance Status of 0 or 1 at both the screening and baseline visits;
6. Life expectancy ≥12 weeks;
7. Adequate laboratory parameters during screening as evidenced by:

   * Absolute neutrophil count ≥1.5×109/L (1500/mm3)
   * Platelets ≥100×109/L (100,000/mm3)
   * Hemoglobin (Hgb) ≥9.0 g/dL (90 g/L)
   * Albumin levels ≥2.8 g/dL
   * Total bilirubin ≤1.5 times the upper limit of normal (× ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN; for subjects with liver metastases, ALT and AST ≤5× ULN
   * Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min (using Cockcroft-Gault equation)
8. Female subjects agree not to be pregnant or lactating from beginning of the study screening to 3 months after receiving the last treatment:

   * Both men and women of reproductive potential are willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy
   * A highly effective method of contraception is defined as one that results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly
9. Willing and able to comply with clinic visits and study-related procedures;
10. Provide signed informed consent.

Exclusion Criteria

Subjects who fulfill any of the following criteria at screening will be ineligible to participate in this study:

1. Known history of hypersensitivity to any components of the SHR-1316 product;
2. Any investigational or concurrent cancer therapy (including surgery, radiotherapy, immunotherapy, hormone therapy, or target therapy), administered within 4 weeks or 5 half-lives, whichever is longer, before the first dose of SHR-1316; or within 6 weeks in the case of certain therapies (e.g., extensive radiotherapy, major surgery, mitomycin C and nitrosoureas). Any such, prior systemic therapy needs to be outside of five half-lives, unless discussed and explained with the sponsor. Any AEs from prior therapy must have returned to ≤ Grade 1 CTCAE level;
3. Subjects with active, known, or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid patients with a history of Grave's disease (subjects with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study drug), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
4. Active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease. Prior treated brain or meningeal metastases must be clinically stable (MRI) for at least 8 weeks and off immunosuppressive doses of systemic steroids (<10 mg/day prednisone or equivalent) for at least 4 weeks before study drug administration;
5. Clinically significant cardiovascular condition, including: (1) history of congestive heart failure (NYHA Class >2), (2) history of unstable angina, (3) myocardial infarction within the past 12 months, or (4) history of supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
6. History or presence of an abnormal ECG that, in the investigator's opinion, is clinically meaningful:

   • For example, a screening QTcF interval that is prolonged (>450 milliseconds [msec] in males; >470 msec in females).
7. Active infection or an unexplained fever >38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled);
8. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or any active systemic viral infection requiring therapy (e.g., hepatitis B or C);
9. Any other medical (e.g., pulmonary, metabolic, congenital, endocrinal or CNS disease, etc.), psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare or ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 3 weeks
  Incidence of treatment-related AEs
Laboratory parameters | Up to 3 weeks
  Incidence of clinically significant laboratory abnormalities
Vital sign values | Up to 3 weeks
  Incidence of clinically significant vital sign abnormalities
ECG values | Up to 3 weeks
  Incidence of clinically significant ECG abnormalities
Dose-limiting toxicities (DLTs) | Up to 3 weeks
  Number of participants with DLTs

SECONDARY OUTCOMES:
Tmax | Cycle 1 Day 1 (pre-dose and 5 min, 1 hr, 2 hr, and 6 hr post-dose), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22; Day 1 from Cycle 2 onwards (pre-dose and 5-min post-dose)
  Time to maximum plasma concentration
Cmax | Cycle 1 Day 1 (pre-dose and 5 min, 1 hr, 2 hr, and 6 hr post-dose), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22; Day 1 from Cycle 2 onwards (pre-dose and 5-min post-dose)
  Maximum plasma drug concentration
AUC | Cycle 1 Day 1 (pre-dose and 5 min, 1 hr, 2 hr, and 6 hr post-dose), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22; Day 1 from Cycle 2 onwards (pre-dose and 5-min post-dose)
  Area under the time-concentration curve
t1/2 | Cycle 1 Day 1 (pre-dose and 5 min, 1 hr, 2 hr, and 6 hr post-dose), Day 2, Day 3, Day 4, Day 8, Day 15, Day 22; Day 1 from Cycle 2 onwards (pre-dose and 5-min post-dose)
  Observed terminal half-life
Receptor occupancy | Cycle 1 Day 1 (pre-dose, 1 hr post-dose); Cycle 1 Day 4; Cycle 1 Day 8; Cycle 1 Day 15; Cycle 2 Day 1; Cycle 3 Day 1
  PD-1 receptor occupancy in blood
Immunogenicity | Cycle 1 Day 1 (pre-dose), Cycle 1 Day 8, Cycle 1 Day 15; pre-dose on Day 1 of Cycle 2 onwards
  Incidence of anti-SHR-1316 antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No